CLINICAL TRIAL: NCT06178614
Title: A Phase 1 Study of JNJ-87890387, an Ectonucleotide Pyrophosphatase/Phosphodiesterase Family Member 3 (ENPP3) x CD3 Bispecific Antibody, for Advanced Solid Tumors
Brief Title: A Study of JNJ-87890387 for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109339; 87890387STM1001 (Other: Janssen Research & Development, LLC); 2023-505358-16-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-87890387 (Experimental): In Part 1 (Dose escalation) participants will receive JNJ-87890387. The dose will be escalated sequentially until the recommended phase 2 dose (RP2D) regimen(s) have been identified. In Part 2 (Dose expansion), participants will receive JNJ-87890387 at the RP2D regimen(s) determined in Part 1.
  Interventions: Drug: JNJ-87890387

INTERVENTIONS:
Drug: JNJ-87890387 — JNJ-87890387 will be administered.

SUMMARY:
The purpose of this study is to determine safety and recommended phase 2 dose(s) (RP2Ds) of JNJ-87890387 and to determine the safety of JNJ-87890387 at the RP2D(s).

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed, metastatic, or unresectable solid tumor of one of the following types: a) Renal cell cancer (RCC)-clear cell or papillary carcinoma; b) Endometrioid ovarian cancer c) Endometrioid uterine carcinoma; d) Colorectal adenocarcinoma (CRC); e) Lung adenocarcinoma
* Have measurable or evaluable disease: Part 1- Either measurable or evaluable disease; Part 2- At least 1 measurable lesion per RECIST v1.1. Participants with ovarian cancer without a measurable lesion must have disease evaluable per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) or have cancer antigen (CA) 125 greater than (>) 2*upper limit of normal (ULN) during screening
* All participants in Part 1 and Part 2 must consent to provide an archived tumor tissue sample at screening
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at screening
* Be willing and able to adhere to the lifestyle restrictions specified in this protocol.

Exclusion Criteria:

* Active Central Nervous System (CNS) involvement with the exception of locally treated brain metastases that are clinically stable and asymptomatic for > 2 weeks and who are off or receiving low-dose corticosteroid treatment (less than or equal to [<=]10 milligrams [mg] prednisone or equivalent) for at least 2 weeks prior to start of study treatment
* Toxicity from prior anticancer therapy that has not resolved to Grade <=1 (except alopecia, vitiligo, Grade <=2 peripheral neuropathy, or endocrinopathies that are stable on hormone replacement)
* History of Grade greater than or equal to (>=) 2 immune-related AE(s) with prior immunotherapy that led to discontinuation of previous immunotherapy with the exception of Grade 2 and Grade 3 immune-related AEs that responded to treatment and that did not recur following rechallenge. Endocrinopathies that are stable on hormone replacement therapy or that have resolved are allowed.
* History of solid organ or hematologic stem cell transplantation
* Any episode of partial or complete bowel obstruction requiring hospitalization within 30 days prior to first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2027-03-16 (Estimated); Study Completion 2029-02-07 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose Limiting Toxicity (DLTs) | Up to first 21 days after administration of the first full treatment dose
  Number of participants with DLTs will be reported. The DLTs are adverse events including certain high grade non-hematologic or hematologic toxicities, or toxicities meeting other specific criteria.
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) by Severity | Up to 2 years 9 months
  An AE is any untoward medical occurrence in a clinical study participant administered an investigational or non-investigational product and it does not necessarily have a causal relationship with the investigational product. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 with the exception of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome events (ICANS), which will be graded by American Society for Transplantation and Cellular Therapy (ASTCT) guidelines. Severity scale ranges from grade 1 (mild) to grade 5 (death). Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to adverse event.

SECONDARY OUTCOMES:
Part 1 and Part 2: Serum Concentration of JNJ-87890387 | Up to 2 years 9 months
  Serum concentration of JNJ-87890387 will be reported.
Part 1 and Part 2: Maximum Observed Serum Concentration (Cmax) of JNJ-87890387 | Up to 2 years 9 months
  Cmax is defined as maximum observed serum concentration of JNJ-87890387.
Part 1 and Part 2: Time to Reach Maximum Observed Serum Concentration (Tmax) of JNJ-87890387 | Up to 2 years 9 months
  Tmax is defined as the time to reach maximum observed serum concentration of JNJ-87890387.
Part 1 and Part 2: Area Under the Curve from Time t1 to Time t2 (AUC[t1-t2]) of JNJ-87890387 | Up to 2 years 9 months
  AUC(t1-t2) is defined as area under the serum concentration versus time curve from time t1 to time t2 of JNJ-87890387.
Part 1 and Part 2: Area Under the Curve from Time Zero to Time tau (AUC[0-tau]) of JNJ-87890387 | Up to 2 years 9 months
  AUC(0-tau) is defined as area under the serum concentration versus time curve from time 0 to time tau of JNJ-87890387.
Part 1 and Part 2: Minimum Observed Serum Concentration (Cmin) of JNJ-87890387 | Up to 2 years 9 months
  Cmin is defined as the minimum observed serum concentration of JNJ-87890387.
Part 1 and Part 2: Accumulation Ratio of JNJ-87890387 | Up to 2 years 9 months
  Accumulation ratio of JNJ-87890387 will be reported. The AR is the accumulation ratio calculated as Cmax or AUC after multiple doses divided by Cmax or AUC after the first dose, respectively.
Part 1 and Part 2: Number of Participants with Presence of Anti-JNJ-87890387 Antibodies | Up to 2 years 9 months
  Number of participants with presence of anti-JNJ-87890387 antibodies will be reported.
Part 1 and Part 2: Objective Response Rate (ORR) | Up to 2 years 9 months
  ORR is defined as the percentage of participants with a best response of complete response or partial response according to Response Evaluation Criteria in Solid Tumors (RECIST) maintained for at least 4 weeks.
Part 1 and Part 2: Duration of Response (DOR) | Up to 2 years 9 months
  DOR is defined as the duration from the date of initial documentation of a response to the date of first documented evidence of disease progression according to RECIST v. 1.1, or death due to any cause, whichever occurs first.

OTHER OUTCOMES:
Part 1 and Part 2: Time to Response (TTR) | Up to 2 years 9 months
  TTR is defined for the responders as the time from the date of the first dose of JNJ-87890387 to the date of the first documented response.
Part 1 and Part 2: Cancer Antigen (CA) 125 Response Rate | Up to 2 years 9 months
  CA 125 response rate is defined as the proportion of participants with ovarian cancer who achieved a partial response or complete response according to the Gynecologic Cancer Intergroup (GCIG) response criteria for CA 125, maintained for at least 4 weeks. A CA 125 response is defined as at least 50 percentage (%) reduction in CA 125 levels from a pretreatment sample which must be confirmed and maintained for at least 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- United States (2):
  - Start Midwest, Grand Rapids, Michigan
  - Sarah Cannon Research Institute, Nashville, Tennessee
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Spain (2):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency